CLINICAL TRIAL: NCT03315611
Title: Study to Assess the Effect of "Eucerin AtopiControl" on Dermal Symptoms in Patients With Atopic Dermatitis After Challenges With Grass Pollen in the Fraunhofer Allergen Challenge Chamber
Brief Title: Study to Assess the Effect of "Eucerin AtopiControl" on Dermal Symptoms in Patients With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-09 Neurop 2
Record Dates: First submitted 2017-10-02; First posted 2017-10-20 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2017-10

CONDITIONS: Atopic Dermatitis; Allergy Pollen
MeSH Terms: conditions — Dermatitis, Atopic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Intervention Model Description: The working hypothesis fo this study is, that local treatment with 'Eucerin AtopiControl Lotion' and 'Eucerin AtopiControl Gesichtscreme' compared to no treatment signifixantly reduces the increase of SCORAD that is elicited during challenge in an environmental challenge chamber (ECC) with grass pollen.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AD, sensitized, treated (Active Comparator): Allergen challenge chamber and Treatment for 12 day with 'Eucerin AtopiControl Lotion' (for the body) and 'Eucerin AtopiControl facial cream' (for the face): 1,2 g twice daily.
  Interventions: Drug: 'Eucerin AtopiControl Lotion' (for the body); Other: Allergen challenge chamber
- AD, not sensitized, not treated (Experimental): Allergen challenge chamber
  Interventions: Other: Allergen challenge chamber
- AD, sensitized, not treated (Experimental): Allergen challenge chamber
  Interventions: Other: Allergen challenge chamber

INTERVENTIONS:
Drug: 'Eucerin AtopiControl Lotion' (for the body) — Treatment with Eucerin AtopiControl Lotion
  Other Names: 'Eucerin AtopiControl facial cream' (for the face); Two 4h-challenges with grass pollen on two consecutive days
  Arms: AD, sensitized, treated
Other: Allergen challenge chamber — Exposure to Dactylis glomerata pollen in an environmental challenge chamber

SUMMARY:
The objective of this study is to assess the effect of 'Eucerin AtopiControl LOTION' and 'Eucerin AtopiControl facial cream' on dermal symptoms in patients with Atopic Dermatitis (AD) after two 4 h challenges with grass pollen on two consecutive days. In addition, this clinical study with exposure of Dactyls glomerate-sensitized Patients with AD shall be used to compare the skin response with AD Patients not-sensitized to Dactylis glomerata to understand the specificity of the grass pollen exposure.

DETAILED DESCRIPTION:
After the screening assessments the subject's whole skin will be treated for a period of 12 days with either 'Eucerin AtopiControl LOTION' or 'Eucerin AtopiControl facial cream' or will receive no treatment until Day 1 of the study. All patients will be challenged for 4 hours on two consecutive days (Day1 and 2) with 4000 pollen grains/m³ of Dactylis glomerata pollen. In this study approximately 9 subjects will be placed in the Environmental Exposure Chamber (ECC) at a time. At screening a blood sample will be taken for determination mutations of genes encoding for skin barrier proteins (e.g. filaggrin mutation). At day 1 and day 5 blood samples (serum) will be taken for biomarker assessments and lymphocyte proliferation assays (peripheral blood). The severity of atopic dermatitis will be rated (blinded observer, trained dermatologist) applying the 'SCORing Atopic Dermatitis (SCORAD) index, the objective SCORAD, local SCORAD and Investigator Global assessment (IGA). Assessment of itch and sleeplessness referring to the past 24 hous will be done by a blinded observer on each day including baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* Women will be considered for inclusion if they are: not pregnant, as confirmed by pregnancy test (see flow chart) and not nursing.

Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit). Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after the last pollen challenge -, implants, injectables, combined oral contraceptives, hormonal Intra Uterine Devices (IUD) or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).

* For patient groups 1 and 2: Positive Immunglobulin E (IgE) level for Dactylis glomerata of at least ImmunoCAP fluoroenzyme immunoassay (CAP FEIA) class 3 at screening or within the last 12 months.
* atopic dermatitis fulfilling the United Kingdom (UK) criteria of AD
* SCORAD index between 20 and 50 points.
* Forced expiratory Volume in 1 second (FEV1) ≥ 80% pred. at screening.
* Smokers or non-smokers
* Applicable only for patients of the control group: No IgE-sensitization to grass pollen (including Dactylis glomerata)

Exclusion Criteria:

* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease.
* Asthma other than mild asthma which is treated with short acting beta-2-agonists only and which is controlled according to the current GINA (Global Initiative for Asthma) guidelines
* Clinically relevant abnormalities in hematology or blood chemistry at screening.
* Positive Human Immunodeficiency Virus Antibody (HIV-1/2Ab), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HCV-Ab) test at screening.
* Treatment with medication that might interfere with rescue medication for anaphylactic reactions (e.g. beta blocker).
* Topical steroid treatment of air exposed skin (wash out phase: 2 weeks)
* Topical calcineurin inhibitor treatment of air exposed skin (wash out phase: 2 weeks)
* Ultraviolet (UV) radiation treatment (wash out phase: 4 weeks)
* Systemic immunosuppression treatment (steroids, cyclosporine, azathioprine, Mycophenolate Mofetil (MMF); wash out phase: 4 weeks)
* Treatment with antihistamines (wash out phase: 1 week)
* Specific immunotherapy (SIT) with grass pollen allergens within the last 5 years
* Diastolic blood pressure above 95 mmHg.
* Febrile illness within 2 weeks prior to screening.
* Alcohol or drug abuse within 12 month prior to screening.
* Regular daily consumption of more than 1 liter of usual beer or the equivalent quantity of approximately 40 g of alcohol in another form.
* Participation in another clinical trial 30 days prior to enrolment.
* Risk of non-compliance with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
SCORAD Day 3 | Day 3: pre- 4 hour-challenge with grass pollen and post-4 hour-challenge with grass pollen
  Difference of change in objective SCORAD in treated versus untreated patients

SECONDARY OUTCOMES:
SCORAD Day 1,2,4,5 | Day 1,2,4,5: pre- 4 hour -challenge with grass pollen and post-4 hour-challenge with grass pollen
  Difference of change in objective SCORAD in treated versus untreated patients

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Principal Investigator — The Fraunhofer-Gesellschaft
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany